CLINICAL TRIAL: NCT01270945
Title: Phase II Open Label,Randomized Study of the Safety, Pharmacokinetics, and Preliminary Efficacy of an Anti-Inflammatory Therapeutic Antibody(CV-18C3)in Reducing Restenosis in Patients Undergoing Percutaneous Femoro-popliteal Revascularization.
Brief Title: Safety and Preliminary Efficacy Study of an Anti-inflammatory Therapeutic Antibody in Reducing Restenosis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-PT017
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Patients Undergoing Repeat Peripheral Artery Revascularization
MeSH Terms: interventions — bermekimab; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CV-18C3 and standard of care (Experimental): CV-18C3 and standard of care
  Interventions: Drug: CV-18C3; Procedure: Standard of Care
- standard of care (Active Comparator): Percutaneous revascularization
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Drug: CV-18C3 — 3.75mg/kg given IV for a period of 6 weeks, followed by subcutaneous administration
  Arms: CV-18C3 and standard of care
Procedure: Standard of Care

SUMMARY:
The purpose of this study is to determine if CV-18C3 will reduce the rate of restenosis or the time to restenosis in patients undergoing repeat peripheral artery revascularization versus controls randomized to standard of care.

DETAILED DESCRIPTION:
Restenosis of peripheral artery lesions remains a challenging problem to overcome after percutaneous revascularization of atherosclerotic disease in the femoropopliteal arterial system. Rates of restenosis are as high as 60% after a year. Treatment options include medical therapy, angioplasty, arthrectomy and stent placement. The heterogeneity of disease between patients, variable length of target lesions and presence of unpredictable physical forces requires individualized treatment plans.

Vascular response to injury appears to play an important role in the development of restenosis. IL-1α is a potent inflammatory cytokine that plays a central role in vascular inflammation and vascular smooth muscle proliferation--both in acute and chronic injury. CV-18C3 antagonizes the biologic activity of IL-1α and is theorized to prevent the early IL-1α mediated inflammation that leads to vascular smooth muscle hypertrophy and restenosis, as well as the late IL-1α mediated atherosclerotic plaque formation.

ELIGIBILITY:
Inclusion Criteria:

* Have suspected superficial femoro-popliteal artery occlusion due to lower extremity pain with exercise or at rest and are undergoing a planned arteriogram.
* Subjects will be randomized after angiographic evidence of qualifying lesion

Exclusion Criteria:

* Acute critical limb ischemia
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-06-30 (Actual); Primary Completion 2013-09-30 (Actual); Study Completion 2014-04-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of CV-18C3 | 1 year
  adverse events, vitals signs, physical examination results and clinical laboratory values

SECONDARY OUTCOMES:
Time to restenosis and restenosis rates compared between CV-18C3 and controls | 1 year
  Efficacy determination will be derived from observed rates of target vessel occlusion, time to occlusion, incidence of target vessel revascularization procedures and incidence of major adverse cardiovascular events (MACE). ABI measurements and quality of life questionnaire scores will also be collected. Treated subjects will be compared to those randomized to no treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hosam El-Sayed, M.D., Ph.D., Principal Investigator — Methodist Cardiovascular Surgery Associates
Locations (8):
- United States (8):
  - Sutter Heart & Vascular Institute, Sacramento, California
  - JFK Medical Center, Atlantis, Florida
  - River City Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Mediquest Research Group, Ocala, Florida
  - John D. Archbold Memorial Hospital, Thomasville, Georgia
  - Univeristy of Cincinnati University Hospital, Cincinnati, Ohio
  - Methodist Hospital, Houston, Texas

REFERENCES:
- [Derived] El Sayed H, Kerensky R, Stecher M, Mohanty P, Davies M. A randomized phase II study of Xilonix, a targeted therapy against interleukin 1alpha, for the prevention of superficial femoral artery restenosis after percutaneous revascularization. J Vasc Surg. 2016 Jan;63(1):133-41.e1. doi: 10.1016/j.jvs.2015.08.069. Epub 2015 Oct 1. PMID 26433546